CLINICAL TRIAL: NCT04339673
Title: Comparison of the Efficacy of Different Treatment Modalities in Masseteric Myofascial Pain: Masseteric Nerve Block, Local Anesthetic Injection and Dry-needling
Brief Title: Is Masseteric Nerve Block Effective in Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Fatih TASKESEN, Head of Dept. Oral and Maxillofacial Surgery, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 135162
Record Dates: First submitted 2020-04-02; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Myofascial Pain - Dysfunction Syndrome of TMJ; Myofascial Trigger Point Pain; Local Anesthesia
Keywords: pain; injections; anesthetics
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes; Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: randomized parallel controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MNB- masseteric nerve block (Active Comparator): masseteric nerve block with local anesthesia lidocaine single app.
  Interventions: Procedure: masseteric nerve block
- LA -trigger point injection with local anesthetic (Active Comparator): local anesthetic injections on trigger points in masseter
  Interventions: Procedure: trigger point injection
- DN-dry needling (Placebo Comparator): dren needling to masseter
  Interventions: Procedure: dry needling

INTERVENTIONS:
Procedure: masseteric nerve block — regional bloc of masseter
  Arms: MNB- masseteric nerve block
Procedure: trigger point injection — trigger point injection with local anesthetic
  Arms: LA -trigger point injection with local anesthetic
Procedure: dry needling — needling with acupuncture needles of trigger points in masseter
  Arms: DN-dry needling

SUMMARY:
The aim of the present study was to compare the efficacy of three different treatment methods in the management of myofascial pain: masseteric nerve block (MN), trigger point injection(TrP) with local anesthetic (LA) and dry needling (DN).Study Design: 45 subjects aged 18-54 years were randomly assigned to the MN group (n= 15), LA group (n=15) and DN group (n=15).

DETAILED DESCRIPTION:
The study sample consisted 45 patients with masseter muscle originated myofascial pain, were selected in accordance with the following criteria:

Patients were grouped according to the treatment they received: dry-needling (DN), TrP injections with local anesthetic (LA) and masseteric nerve block (MNB). Localization of the masseteric trigger points (MTPs) was based on clinician's sense and patients' expressions of pain. Local twitch response was not observable in all case. This procedure was completed by using digital palpation (1.5 Kg), and the clinical examiner's palpation was calibrated using a pressure algometer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of myofascial pain.
* Presence of at least one trigger point in masseter muscle.

Exclusion Criteria:

* Generalized muscle disorders.
* Hypersensitivity to local anesthetics.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
The Rate of Pain on Function (PoF) assessed by Numerical pain Scale (NRS) | before the injections (T0, Baseline)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The Rate of Pain on Function (PoF) assessed by Numerical pain Scale (NRS) | At 1st week (t1)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The Rate of Pain on Function (PoF) assessed by Numerical pain Scale (NRS) | At 4th week (t2)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The Rate of Pain on Function (PoF) assessed by Numerical pain Scale (NRS) | At 12th week (t3)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)

SECONDARY OUTCOMES:
The Rate of Pain Intensity on Palpation (PoP) | before the injections (T0, Baseline)
  Patients rated their pain intensity on masseter muscle by a 4-point Likert-type scale (0 = no pain, 3 = as worst pain imaginable) while a calibrated examiner palpating their masseter muscle.
The Rate of Pain Intensity on Palpation (PoP) | At 1st week (t1)
  Patients rated their pain intensity on masseter muscle by a 4-point Likert-type scale (0 = no pain, 3 = as worst pain imaginable) while a calibrated examiner palpating their masseter muscle.
The Rate of Pain Intensity on Palpation (PoP) | At 4th week (t2)
  Patients rated their pain intensity on masseter muscle by a 4-point Likert-type scale (0 = no pain, 3 = as worst pain imaginable) while a calibrated examiner palpating their masseter muscle.
The Rate of Pain Intensity on Palpation (PoP) | At 12th week (t3)
  Patients rated their pain intensity on masseter muscle by a 4-point Likert-type scale (0 = no pain, 3 = as worst pain imaginable) while a calibrated examiner palpating their masseter muscle.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | before the injections (T0, Baseline)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain in masseter muscle. Three measurements were performed, and their average is recorded.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | At 1st week (t1)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain in masseter muscle. Three measurements were performed, and their average is recorded.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | At 4th week (t2)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain in masseter muscle. Three measurements were performed, and their average is recorded.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | At 12th week (t3)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain in masseter muscle. Three measurements were performed, and their average is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Ağiz Ve Diş Sağlığı Egt Araş Hastanesi, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venancio Rde A, Alencar FG Jr, Zamperini C. Botulinum toxin, lidocaine, and dry-needling injections in patients with myofascial pain and headaches. Cranio. 2009 Jan;27(1):46-53. doi: 10.1179/crn.2009.008. PMID 19241799
- [Result] Quek SY, Subramanian G, Patel J, Ananthan S, Zagury JG, Khan J. Efficacy of regional nerve block in management of myofascial pain of masseteric origin. Cranio. 2015 Oct;33(4):285-90. doi: 10.1080/08869634.2015.1097300. Epub 2015 Dec 29. PMID 26715419

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04339673/Prot_SAP_000.pdf